CLINICAL TRIAL: NCT00986869
Title: Study of the Safety of Flexible Bronchoscopy in Patients With Pulmonary Hypertension
Brief Title: The Safety of Flexible Bronchoscopy in Patients With Pulmonary Hypertension
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 128-09
Record Dates: First submitted 2009-09-23; First posted 2009-09-30 (Estimated); Last update posted 2012-03-16 (Estimated); Status verified 2012-03

CONDITIONS: Pulmonary Hypertension
Keywords: Safety; Bronchoscopy; Pulmonary; Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary; Hypertension

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- echocardiogram: All the patients will undergo a Doppler echocardiogram in the day of the bronchoscopy after the bronchoscopy
  Interventions: Procedure: Doppler echocardiogram

INTERVENTIONS:
Procedure: Doppler echocardiogram — All the patients will undergo a Doppler echocardiogram in the day of the bronchoscopy after the bronchoscopy

SUMMARY:
Background

Flexible bronchoscopy (FB) is one of the most common invasive procedures performed by pulmonologists (1) . Typically performed under topical anesthesia and conscious sedation, the procedure is considered to be safe, effective and well tolerated in patients with a wide variety of pulmonary diseases (2). Complications associated with the procedure are rare and studies have estimated an incidence of 0.5-4% (3) The most commonly recognized complications include hypoxia, bleeding, bronchospasm, cardiac dysrhythmias, pneumothorax, and vagal reactions (4). Several conditions increase the risk of complications including pre-existent hypoxemia, use of mechanical ventilation, uremia, profound thrombocytopenia, coagulopathy and pulmonary hypertension (PH) (5). Although previous reports suggest that transbronchial biopsies increase the risk for hemorrhage in this population, data are is limited to survey analyses and isolated reports. Recently Guzman et al. reported a retrospective analysis about the safety of FB in PH. (6) They found that FB can be performed safely in patients with mild and moderate PH. However, the study was small and retrospective analysis. Furthermore, there is no consensus regarding levels of pulmonary artery pressure (PAP) considered to be safe for invasive diagnostic interventions such as TBLB or transbronchial needle aspiration.

Objective

To assess the safety of FB in patients with PH and to study the occurrence of complications associated with different diagnostic bronchoscopic procedures.

DETAILED DESCRIPTION:
The Safety of Flexible Bronchoscopy in Patients with Pulmonary Hypertension

1Pulmonary department and 2Devision of Cardiology Affiliated with Sackler Faculty of Medicine, Tel Aviv University, Tel Aviv, Israel; Meir Medical Center, Kfar Saba, Israel

Background

Flexible bronchoscopy (FB) is one of the most common invasive procedures performed by pulmonologists (1) . Typically performed under topical anesthesia and conscious sedation, the procedure is considered to be safe, effective and well tolerated in patients with a wide variety of pulmonary diseases (2). Complications associated with the procedure are rare and studies have estimated an incidence of 0.5-4% (3) The most commonly recognized complications include hypoxia, bleeding, bronchospasm, cardiac dysrhythmias, pneumothorax, and vagal reactions (4). Several conditions increase the risk of complications including pre-existent hypoxemia, use of mechanical ventilation, uremia, profound thrombocytopenia, coagulopathy and pulmonary hypertension (PH) (5). Although previous reports suggest that transbronchial biopsies increase the risk for hemorrhage in this population, data are is limited to survey analyses and isolated reports. Recently Guzman et al. reported a retrospective analysis about the safety of FB in PH. (6) They found that FB can be performed safely in patients with mild and moderate PH. However, the study was small and retrospective analysis. Furthermore, there is no consensus regarding levels of pulmonary artery pressure (PAP) considered to be safe for invasive diagnostic interventions such as TBLB or transbronchial needle aspiration.

Objective To assess the safety of FB in patients with PH and to study the occurrence of complications associated with different diagnostic bronchoscopic procedures.

Materials and Methods Study Population 100 patients that will undergo a bronchoscopy according to the regular indications during the study period (12 months) will be eligible for the study.

Criteria for exclusion Exclusion criteria will be age under 18 years and patients who are unable to obtain informed consent. Patients with known severe pulmonary hypertension (PAP above 70 mmHg) will be exclude from the study.

Procedural Conduct All procedures will be performing in the bronchoscopy suite of the Pulmonary Department in Meir Medical center. Fluoroscopy will be available for all procedures. FB will be performed by a training pulmonary physician that will be blinded to the echocardiograpgic findings. Oxygen will be administered to all patients to ensure SpO2 >90% prior to the introduction of the bronchoscope. Continuous pulse oximetry, electrocardiogram and noninvasive blood pressure monitoring will be obtained throughout the procedure. Sedation will be achieved using midazolam. Topical anesthesia (was) will be obtained using 2% lidocaine.

Study Subjects All the patients will undergo a Doppler echocardiogram in the day of the bronchoscopy after the bronchoscopy. The diagnosis of PH will define as (1) mean PAP (mPAP) >25 mm Hg measured by right heart catheterization (RHC), or (2) right ventricular systolic pressure (RVSP) >40 mm Hg estimated by Doppler echocardiography.

PAP will be calculated as the sum of tricuspid regurgitation gradient and estimated right atrial pressure, provided there is no increase in pulmonic valve flow velocity .Maximal tricuspid regurgitation velocity (taken from all available views) will be measured by continuous wave Doppler echocardiography to evaluate the pressure gradient from the right ventricle to the right atrium. Right atrial pressure will be estimated on the basis of inferior vena cava (IVC) size and inspiratory collapse (7,8).

Data Collection Data will be collected from all patients including baseline characteristics of age, sex, medications and electrocardiogram. Blood tests including blood count, indication for bronchoscopy, duration and bronchoscopic procedures. All echocardiogram findings will be collected by physicians that will be blinded to the bronchoscpoic details.

Outcome Measures The primary outcome will be the incidence of complications after FB. Complications will define as hypoxemia (SpO2 <90% and need of supplemental oxygen within 30 min of a completed procedure), hypotension (mean arterial pressure <60 mm Hg or systolic blood pressure <90 mm Hg for more than 5 min and/or need for administration of intravenous solution or vasopressors), cardiac dysrhythmias (new onset of arrhythmia or worsening of underlying arrhythmia that caused hemodynamic instability and/or required urgent intervention), bleeding, and death.

The amount of bleeding will be estimated as: no bleeding - minimal bleeding that does not require suctioning; mild bleeding - the need to continually suction the airways; moderate bleeding - the need to wedge FB in the segment involved; severe bleeding - the need for additional interventions or transfusion.

Statistical Analysis Results will express as the mean ± SD for continuous variables. Qualitative data will express as the percentage of patients with a 95% confidence interval. Nominal variables will be compared with Pearson's 2 or Fisher's exact test. Continuous outcome variables will be compared using Student's t test or rank-sum tests as appropriate. Statistical significance will be defined as p < 0.05.

Statistical analysis will be performed using a statistical software package (SPSS, version 13.0; SPSS Inc., Chicago, Ill., USA).

ELIGIBILITY:
Inclusion Criteria:

* All patients that will undergo a bronchoscopy according to the regular indications during the study period (12 months) will be eligible for the study.

Exclusion Criteria:

* Exclusion criteria will be age under 18 years and patients who are unable to obtain informed consent.
* Patients with known severe pulmonary hypertension (PAP above 70 mmHg) will be exclude from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients that will undergo a bronchoscopy according to the regular indications during the study period (12 months) will be eligible for the study.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2009-09; Primary Completion 2012-08 (Estimated); Study Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
The primary outcome will be the incidence of complications after FB. Complications will define as hypoxemia, hypotension cardiac dysrhythmias, bleeding, and death. | one year

CONTACTS AND LOCATIONS:
Overall Officials: Michael kutuk, Study Chair — Meir Medical Center
Locations (1):
- Meir Medical Center, Kfar Saba, Israel

REFERENCES:
- [Background] Colt HG, Prakash UBS, Offord KP: Bronchoscopy in North America: survey by the American Association for Bronchology, 1999. J Bronchol 2000;7:8-25.
- [Background] Ernst A, Silvestri GA, Johnstone D; American College of Chest Physicians. Interventional pulmonary procedures: Guidelines from the American College of Chest Physicians. Chest. 2003 May;123(5):1693-717. doi: 10.1378/chest.123.5.1693. No abstract available. PMID 12740291
- [Background] Pue CA, Pacht ER. Complications of fiberoptic bronchoscopy at a university hospital. Chest. 1995 Feb;107(2):430-2. doi: 10.1378/chest.107.2.430. PMID 7842773
- [Background] Pereira W Jr, Kovnat DM, Snider GL. A prospective cooperative study of complications following flexible fiberoptic bronchoscopy. Chest. 1978 Jun;73(6):813-6. doi: 10.1378/chest.73.6.813. PMID 657853
- [Background] Guidelines for fiberoptic bronchoscopy in adults. American Thoracic Society. Medical Section of the American Lung Association. Am Rev Respir Dis. 1987 Oct;136(4):1066. doi: 10.1164/ajrccm/136.4.1066. No abstract available. PMID 3662229